CLINICAL TRIAL: NCT02191761
Title: Phase1, Open-Label, Dose Escalation, Dose-Finding Study Evaluating the Safety and Pharmacokinetics of SM04755 in Subjects With Advanced Colorectal, Gastric, Hepatic, or Pancreatic Cancer
Brief Title: Safety and Pharmacokinetics of SM04755 in Subjects With Advanced Colorectal, Gastric, Hepatic, or Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM04755-ONC-01
Record Dates: First submitted 2014-06-30; First posted 2014-07-16 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer; Gastric Cancer; Hepatic Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SM04755 (Experimental)
  Interventions: Drug: SM04755

INTERVENTIONS:
Drug: SM04755 — Escalating Doses

SUMMARY:
This is an open-label, multi-center, dose escalation study in adult subjects with advanced colorectal, gastric, hepatic or pancreatic cancer. The study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of SM04755 administered orally. Upon determination of the maximum tolerated dose (MTD), expansion cohorts may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced colorectal, gastric, hepatic or pancreatic cancer
* Subjects must have recovered from all toxicity associated with previous chemotherapy, targeted therapy, or radiotherapy
* Subjects must meet certain laboratory criteria
* Expected survival > 3months
* Subjects must have no uncontrolled intercurrent illness

Exclusion Criteria:

* Women who are pregnant or lactating, or who are of childbearing potential , and men who do not use a barrier method
* Subjects with significant cardiac issues
* Subjects using certain medications
* Subjects with certain medical conditions
* Subjects with brain metastasis
* Subjects who have recently been enrolled in other experimental clinical trials of investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06-19 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2015-05-20 (Actual)

PRIMARY OUTCOMES:
Determine the MTD | 28 days

SECONDARY OUTCOMES:
Incidence of safety parameters including adverse events, laboratory results, vital signs, electrocardiogram (ECG) findings, Eastern Cooperative Oncology Group (ECOG) performance scores, physical and ophthalmic examination findings | 28 days
Area under the plasma concentration (AUC) Versus Time Curve of SM04755 | 30 days
Characterize the pharmacodynamics (PD) of SM04755 by assessment of its preliminary antitumor activity determined by Response Evaluation Criteria in Solid Tumors (RECIST) | 8 weeks
Maximum Observed Plasma Concentration (Cmax) of SM04755 | 30 Days
Half Life of SM04755 | 30 Days
Volume of Distribution of SM04755 | 30 Days
Time to maximum plasma concentration | 30 Days
Accumulation ratio of SM04755 | 30 Days
Total Clearance of SM04755 after oral administration | 30 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - La Jolla, California
  - Houston, Texas